CLINICAL TRIAL: NCT00597948
Title: Efficacy of a Health Intervention for People With Intellectual Disabilities
Brief Title: Healthy Lifestyles for People With Intellectual Disabilities
Acronym: HLID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Willi Horner-Johnson, Research Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21HD055189-01 (NIH); 1R21HD055189-01 (NIH)
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Mental Retardation; Developmental Disabilities; Intellectual Disabilities
Keywords: mental retardation; downs syndrome; autism; autism spectrum disorder; cerebral palsy; developmental disability; developmental disabilities; intellectual disability; intellectual disabilities; health promotion; disease prevention; physical health; emotional health; behavioral health; mental health; spiritual health; prevention
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Down Syndrome; Autistic Disorder; Autism Spectrum Disorder; Cerebral Palsy; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Workshop Group: Receives Healthy Lifestyles curriculum and subsequent support.
  Interventions: Behavioral: Healthy Lifestyles Curriculum
- 2 (No Intervention): Comparison Group: Does not receive Healthy Lifestyles curriculum and subsequent support.

INTERVENTIONS:
Behavioral: Healthy Lifestyles Curriculum — Three consecutive days of six hours of training comprised of instruction and participant interaction.
  Arms: 1

SUMMARY:
Relatively few health promotion and disease prevention programs have included or targeted people with disabilities, and even fewer have focused on individuals with intellectual disabilities.

The long-term objectives of the Healthy Lifestyles for People with Intellectual Disabilities Study (HLID) are to increase the health of persons with intellectual disabilities by establishing the efficacy of a health promotion program and promoting its adoption. The HLID Study is based in the Center on Community Accessibility (CCA) at Oregon Health & Science University. The mission of CCA is to increase the health and health-related quality of life of persons with disabilities.

A pilot study conducted by CCA has established the effectiveness of the Healthy Lifestyles (HL) intervention among a cross-disability population in increasing health behavior adoption. The specific aim of the HLID Study is to test the efficacy of the HL program specifically with adults with intellectual disabilities.

The HLID Study uses a randomized control study design. The HL intervention will be administered to 75 adults and will compare results to those of an additional 75 adults who receive no intervention. Measurement will include anthropometric assessments to measure impacts on overweight and obesity, as well as self-report measures of healthy behaviors, health status, health care utilization, and secondary conditions. Results will be shared with research participants, presented through professional conferences and newsletters, and published in peer-reviewed journals with the assistance of community partners.

ELIGIBILITY:
Inclusion Criteria:

* Living in Oregon or Southwest Washington
* Ages 18-65 years
* Have mild or moderate mental retardation/developmental disability/intellectual disability as defined by Oregon or Washington state (depending on place of residence) developmental disability service delivery system
* Eligible in Oregon or Washington (depending on place of residence) to receive services for people with mental retardation/developmental/intellectual disability
* Living in the community (i.e., group home, with family/friends, on own with or without support)
* Participant defined health status of excellent, good, or fair
* Participant expressed interest in participation in study
* Participant expressed willingness to be assigned to either Workshop or Control study group

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Health Promoting Lifestyles Profile II | Pre, post, and follow-up

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Pre, post, and follow-up
waist circumference | pre, post, and follow-up
Community Integration Questionnaire | pre, post, and follow-up
Healthy Lifestyles Knowledge Test | pre, post, and follow-up
Starting and Continuing Healthy Behaviors | pre, post, and follow-up
Self-Efficacy and Social Support for Activity for Persons with Intellectual Disabilities | pre, post, follow-up
Living Well with a Disability Evaluation | pre, post, follow-up
General Health Survey | pre, post, follow-up
Healthy Lifestyles Goal Tracking Form | post and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Willi Horner-Johnson, Ph.D., Principal Investigator — Oregon Health and Science University/Center on Community Accessibility
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States